CLINICAL TRIAL: NCT02326259
Title: Evaluation of Progression of Diabetic Retinopathy With Rapid Correction of Hyperglycemia
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 22531
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Disease Progression
MeSH Terms: conditions — Diabetic Retinopathy; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Initiation of treatment of diabetes — Treatment of diabetes according to the standard of care.

SUMMARY:
The investigators are doing this research for two reasons. The first is to see how the retina (back of your eye) changes when your blood sugar is treated with medication for the first time. This will help us better understand the progression of a condition known as Diabetic Retinopathy. The second reason is to provide diabetic blood samples, which will possibly help identify biomarkers for diabetic retinopathy. Biomarkers are things that indicate the presence of a specific condition, and indicate a higher likelihood of developing that condition.

DETAILED DESCRIPTION:
The goal of this research is to conduct a study that investigates (1) how diabetic retinopathy progresses when poorly controlled Type 2 diabetic patients initiate intensive blood sugar control and (2) to determine if there are biomarkers that predict progression of diabetic retinopathy. Typically, the retina is thought to undergo rapid progression of diabetic retinopathy, although this has been poorly characterized in a formal study.

The first goal will be quantified by taking initial photos of the retina with the Pictor Plus hand-held fundus camera, as well as monthly photos (when the patient is scheduled for their endocrinology appointments, throughout a 90 day period). The second goal will be accomplished by testing the patient's blood. There will be an initial blood withdraw, as well as blood withdraws at monthly intervals throughout the same 90 day period as the fundus photos.

This study will help us to understand the pathogenesis of diabetic retinopathy, as well as potentially lead to an improved understanding of progression of diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the endocrinology clinic with a hemoglobin A1c of greater than 12.

Exclusion Criteria:

* Patients with other ocular or systemic conditions, including macular degeneration, uveitis, glaucoma, and autoimmune conditions (Rheumatoid Arthritis, Lupus, and other similar conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being seen in the endocrinology clinic at Temple University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Progression of diabetic retinopathy | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: William J Foster, MD, PhD, Principal Investigator — Temple University; Ajay D Rao, MD, MMSc, FACP, Principal Investigator — Temple University; Raul A DeLa Cadena, MD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States